CLINICAL TRIAL: NCT04875169
Title: A Randomized, Double Blind and Placebo Controlled Phase 3 Study to Evaluate Efficacy and Safety of Oral SHR0302 in Subjects Aged 12 Years and Older With Moderate to Severe Atopic Dermatitis
Brief Title: Evaluate Efficacy and Safety of Oral SHR0302 in Subjects Aged 12 Years and Older With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSJ10333
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Core Treatment Active Experimental: SHR0302 Dose#1 (Experimental): Drug: SHR0302 Oral tablets taken once daily (QD) for 16 weeks
  Interventions: Drug: Core Treatment Active Experimental: SHR0302 Dose#1
- Core Treatment Active Experimental: SHR0302 Dose#2 (Experimental): Drug: SHR0302 Oral tablets taken once daily (QD) for 16 weeks
  Interventions: Drug: Core Treatment Active Experimental: SHR0302 Dose#2
- Core Treatment Placebo Comparator: Placebo (Placebo Comparator): Drug: Placebo Oral tablets taken once daily (QD) for 16 weeks
  Interventions: Drug: Core Treatment Placebo Comparator: Placebo
- Extension Treatment Active Experimental: SHR0302 Dose#1 (Experimental): Drug: SHR0302 Oral tablets taken once daily (QD) for 36 weeks
  Interventions: Drug: Extension Treatment Active Experimental: SHR0302 Dose#1
- Extension Treatment Active Experimental: SHR0302 Dose#2 (Experimental): Drug: SHR0302 Oral tablets taken once daily (QD) for 36 weeks
  Interventions: Drug: Extension Treatment Active Experimental: SHR0302 Dose#2

INTERVENTIONS:
Drug: Core Treatment Active Experimental: SHR0302 Dose#1 — Drug: SHR0302 Oral tablets taken once daily (QD) for 16 weeks
  Arms: Core Treatment Active Experimental: SHR0302 Dose#1
Drug: Core Treatment Active Experimental: SHR0302 Dose#2 — Drug: SHR0302 Oral tablets taken once daily (QD) for 16 weeks
  Arms: Core Treatment Active Experimental: SHR0302 Dose#2
Drug: Core Treatment Placebo Comparator: Placebo — Drug: Placebo Oral tablets taken once daily (QD) for 16 weeks
  Arms: Core Treatment Placebo Comparator: Placebo
Drug: Extension Treatment Active Experimental: SHR0302 Dose#1 — Drug: SHR0302 Oral tablets taken once daily (QD) for 36 weeks
  Arms: Extension Treatment Active Experimental: SHR0302 Dose#1
Drug: Extension Treatment Active Experimental: SHR0302 Dose#2 — Drug: SHR0302 Oral tablets taken once daily (QD) for 36 weeks
  Arms: Extension Treatment Active Experimental: SHR0302 Dose#2

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter Phase 3 study that will enroll approximately 330 subjects aged 12 to 75 years old with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This study consists of a screening period followed by a placebo-controlled treatment period and then an extension treatment period and completed after a follow-up period after the completion of active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects must be at least at ≥12 and ≤75 years of age and body weight ≥40 kg
2. Subject has a diagnosis of atopic dermatitis for at least 1 year.
3. Meets all of the following disease activity criteria: BSA ≥10% of AD involvement. EASI ≥16. IGA ≥3. WI-NRS ≥4
4. Subject has a recent history (within 6 months before the screening visit) of inadequate response or inability to tolerate topical AD treatments (TCS or TCI) or who have required systemic treatments for control of their disease.
5. Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).

Exclusion Criteria:

1. Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, malignancies, current or history of certain infections, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
2. Have received certain treatments that are contraindicated.
3. Subject currently has been diagnosed and has active forms of other inflammatory skin disease (e.g., psoriasis, or lupus erythematosus) that would interfere with the evaluation of atopic dermatitis or response to treatment.
4. Other active non-AD inflammatory skin diseases or conditions affecting skin
5. Subject with active/severe concomitant disease (s)/symptom(s) that requires administering of systemic corticosteroids or otherwise interferes with study participation or requires active frequent monitoring (e.g., unstable chronic asthma).
6. Acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation.
7. Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, malignancies, current or history of certain infections, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
8. Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
9. Subject has any malignancies or has a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
10. Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use contraception.
11. Subject has a previously received systemic JAK inhibitors
12. Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) score of 0/1 at Week 16 | 16 Weeks
  Proportion of subjects achieving Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) and a reduction from baseline of ≥2 points at Week 16.
Eczema Area and Severity Index (EASI 75) at Week 16 | 16 Weeks
  Proportion of subjects achieving at least a 75% improvement in Eczema Area and Severity Index (EASI 75) from baseline at Week 16.

SECONDARY OUTCOMES:
Worst-Itch Numeric Rating Scale (WI-NRS-4)-4 at Week 16 | Week 16
  Proportion of subjects achieving an improvement of Worst-Itch Numeric Rating Scale (WI-NRS) ≥4 from baseline at Week 16
Worst-Itch Numeric Rating Scale (WI-NRS) at Week 1, 4, 8 and 12 | Week 1, 4, 8 and 12
  Proportion of subjects achieving an improvement of WI-NRS ≥4 from baseline at all scheduled visits during placebo-controlled treatment phase other than Week 16.
Time to WI-NRS response | Baseline to Week 16
  Time from baseline to achieve at least 4 points improvement of WI-NRS during placebo-controlled treatment phase.
EASI 75 at Week 1, 4, 8 and 12 | Week 1, 4, 8 and 12
  Proportion of subjects achieving EASI 75 at all scheduled visits during placebo-controlled treatment phase except Week 16.
IGA 0/1 at Week 1, 4, 8 and 12 | Week 1, 4, 8 and 12
  Proportion of subjects achieving IGA0/1 and a reduction from baseline of ≥2 points at all scheduled visits during placebo-controlled treatment phase except Week 16.

OTHER OUTCOMES:
NRS-4 at Week 24, 32, 40, 52 and 56 | All scheduled visits from Week 24 - 56
  Proportion of subjects achieving an improvement of WI-NRS ≥4 from baseline at all scheduled visits during extension treatment phase.
EASI 75 at Week 24, 32, 40, 52 and 56 | All scheduled visits from Week 16 24 - 56
  Proportion of subjects achieving EASI 75 at all scheduled visits during extension treatment phase.
IGA 0/1 at Week 24, 32, 40, 52 and 56 | All scheduled visits from Week 24 - 56
  Proportion of subjects achieving IGA0/1 and a reduction from baseline of ≥2 points at all scheduled visits during extension treatment phase.
EASI 50 and EASI 90 at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Proportion of subjects with ≥50% EASI improvement from baseline (EASI 50) at all scheduled visits.
Change of EASI from baseline at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in the eczema area and severity index (EASI) total score at all scheduled visits. The EASI score ranges from 0.0 to 72.0, can be varied in increments of 0.1, Higher scores indicate greater severity.
SCORAD 50, SCORAD 75 and SCORAD 90 at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  SCORing Atopic Dermatitis (SCORAD). Score of 0-103. Higher scores mean more severe. Proportion of subjects achieving a ≥50%, 75% and 90% improvement in SCORAD (SCORAD 50, SCORAD 75 and SCORAD 90) from baseline at all scheduled visits.
Change of SCORAD from baseline at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in SCORAD at all scheduled visits
Change of BSA from baseline at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in body surface area (BSA) affected at all scheduled visits
Change of IgE from baseline at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in the level of serum IgE in peripheral blood at all scheduled visits.
Change of eosinophils from baseline at Week 1, 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in the level of serum eosinophils in peripheral blood at all scheduled visits.
Change of dermatology life quality index (DLQI) or Children's DLQI (CDLQI) PROs from baseline at Week 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in dermatology life quality index (DLQI) or Children's DLQI (CDLQI) score at all scheduled visits. The DLQI CDLQI consists of questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. This is not a scale. There are no minimum or maximum values. The quality index just captures a subjects perception of the impact of skin disease on different aspects of their health-related quality of life over the last week.
Change of Patient-Oriented Eczema Measure (POEM) from baseline at Week 4, 8, 12, 16, 24, 32, 40, 52 and 56 | Day 1 to Week 56
  Change from baseline in Patient-Oriented Eczema Measure (POEM) at all scheduled visits. 7-item, patient-administered scale that assesses disease severity in children and adults. Subjects respond to questions about the frequency of 7 symptoms (itching, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, and dryness/roughness) over the last week. Response categories include "No days," "1-2 days," "3-4 days," "5-6 days," and "Every day" with corresponding scores of 0, 1, 2, 3, and 4, respectively. Scores range from 0-28 with higher total scores indicating greater disease severity.

CONTACTS AND LOCATIONS:
Locations (52):
- Canada (15):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Dr Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research, Winnipeg, Manitoba
  - CCA Medical Research, Ajax, Ontario
  - SKiN Health, Cobourg, Ontario
  - DermEffects, London, Ontario
  - North York Research Inc., North York, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - York Dermatology, Richmond Hill, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Research Toronto, Toronto, Ontario
  - AvantDerm, Toronto, Ontario
  - XLR8 Clinical Research, Windsor, Ontario
  - Clinique D, Laval, Quebec
- China (37):
  - First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beiing
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhongshan Hospital, Fudan University(Xiamen Branch), Xiamen, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou, Guangdong
  - The First affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hospital for Skin Diseases, Chinese Academy of medical sciences, Nanjing, Jiangsu
  - Jiangsu province people's hospital, Nanjing, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Provincial Hospital of Dermatology, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of jilin university, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Children's Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The first people's hospital of hangzhou, Hangzhou, Zhejiang
  - The fourth hospital affiliated to zhejiang university school of medicine, Yiwu, Zhejiang
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Peking University third hospital, Beijing
  - Peking union medical college hospital, Beijing
  - Children's Hospital Capital Institute of Pediatrics, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - Chongqing Traditional Chinese medicine Hospital, Chongqing
  - First affiliated hospital of chongqing medical university, Chongqing
  - The Southwest Hospital of AMU, Chongqing
  - Zhejiang province People's Hospital, Hangzhou
  - Dermatology hospital of Shanghai, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - The first hospital of China medical university, Shenyang

REFERENCES:
- [Derived] Zhao Y, Gooderham M, Yang B, Wu J, Wu L, Loo WJ, Toth D, Sauder M, Li J, Chen A, Tao X, Lu J, Song Z, Han J, Li H, Li Y, Xu L, Zhang J. Ivarmacitinib for Moderate to Severe Atopic Dermatitis in Adults and Adolescents: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2025 Jul 1;161(7):688-697. doi: 10.1001/jamadermatol.2025.0982. PMID 40305055